CLINICAL TRIAL: NCT06466785
Title: A Phase III, Randomized, Investigator-Blinded, Active-Controlled Study of Efficacy and Safety of Efepoetin Alfa for Treatment of Anemia in Patients With Chronic Kidney Disease on Dialysis
Brief Title: A Phase 3 Study of Efepoetin Alfa for Treatment of Anemia in Patients With Chronic Kidney Disease on Dialysis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Collaborators: PT Kalbe Genexine Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GX-E4-CKD-002
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efepoetin Alfa (GX-E4) (Experimental): Dose: 0.3 mg/0.3 mL, 0.6 mg/0.6 mL and 1 mg/1 mL pre-filled syringe (PFS) solution. The dose of study drug can be varied depending on the level of Hb.
  Frequency: Efepoetin alfa should be administered at 1-week intervals from Day 1 (Visit 2) to Week 28 (Visit 30), but the administration interval may be changed to 1 or 2 weeks from Week 29 (Visit 31) to Week 52 (Visit 54) according to the investigator's judgement.
  Mode of administration: intravenous injection. When the dose of investigational product (IP) is planned on the same day as hemodialysis (HD), the IP should be injected at the end of HD.
  Interventions: Drug: Efepoetin Alfa
- Darbepoetin Alfa (Aranesp®) (Active Comparator): Dose: 20 µg/0.5 mL, 30 µg/0.3 mL, 60 µg/0.3 mL, 100 μg/0.5 mL PFS. The dose of comparator drug can be varied depending on the level of Hb.
  Frequency: Darbepoetin alfa should be administered at 1-week intervals from Day 1 (Visit 2) to Week 28 (Visit 30), but the administration interval may be changed to 1 or 2 weeks from Week 29 (Visit 31) to Week 52 (Visit 54) according to the investigator's judgement.
  Mode of administration: intravenous injection.
  Interventions: Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: Efepoetin Alfa — Efepoetin alfa (Epoetin-Fc fusion protein, GX-E2 or GX-E4,) is a novel long-acting erythropoietin-hybrid fragment crystallizable (Fc) fusion protein developed by Genexine, intended for treatment and maintenance of anemia due to CKD with or without dialysis. Its drug substance is a recombinant form of human EPO and hybrid Fc (hyFc®) fragment consisting of 2 subunits with a total of 411 amino acid residues. Each subunit contains an EPO molecule linked to a hybrid Fc fragment of c terminal of CH2 and CH3 regions from IgG4 and to N-terminal of CH2 region and the hinge sequence from IgD. These 2 subunits are joined by a single disulfide bond at the hinge region of each subunit. Half-life is 138.5-157.9 hours. It is an acidic glycoprotein of about 30 kDa and comprises 165 amino acids and 4 glycans. Circulating EPO exhibits several glycosylation isoforms that differ in electrical charge and biological activity
  Other Names: GX-E4
  Arms: Efepoetin Alfa (GX-E4)
Drug: Darbepoetin Alfa — Darbepoetin alfa is a re-engineered form of erythropoietin containing 5 amino acid changes (N30, T32, V87, N88, T90) resulting in the creation of 2 new sites for N-linked carbohydrate addition. It has a 3-fold longer serum half-life compared to epoetin alpha and epoetin beta. It stimulates erythropoiesis (increases red blood cell levels) by the same mechanism as rHuEpo (binding and activating the Epo receptor) and is used to treat anemia, commonly associated with chronic kidney failure and cancer chemotherapy
  Other Names: Aranesp®
  Arms: Darbepoetin Alfa (Aranesp®)

SUMMARY:
An investigator-blinded, randomized, multicenter, active-controlled Phase III study for the treatment of anemia in patients with CKD on hemodialysis

DETAILED DESCRIPTION:
This is an investigator-blinded, randomized, multicenter, active-controlled Phase III study for the treatment of anemia in patients with CKD on hemodialysis. Eligible patients will be randomized to efepoetin alfa or darbepoetin alfa at a ratio of 2:1. An unblinded team will prepare and administer the study drug at the dosages decided by the blinded Investigator.

The study consists of 3 study periods:

* Screening (up to 28 days before Day 1): subjects in screening will continue treatment with epoetin, methoxy polyethylene glycol-epoetin beta, or darbepoetin alfa as per local standard of care.
* Treatment: subjects will discontinue any prior erythropoietin analogue and will be randomized to switch to efepoetin alfa or darbepoetin alfa in a 2:1 ratio.

The aim of the treatment period is to maintain Hb levels between 10.0 g/dL and 12.0 g/dL. It is recommended that study treatment be administered any time after completion of dialysis if dosing is scheduled on a dialysis day to avoid potential bias on study assessments.

• Follow-up (4 weeks) Phone contacts can be done for follow-up for up to Week 56 or at the time of the last patient's Week 56 visit, whichever is shorter.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females ≥ 18 years old.
2. Patient (or patient's legally acceptable representative) has voluntarily signed and dated an informed consent form (ICF), approved by an Ethics Committee (EC) or institutional review board (IRB), after the nature of the study has been explained and the patient has had the opportunity to ask questions.
3. Patient with stage 5 CKD defined by estimated GFR (eGFR, ≤15 mL/min/1.73m2) on adequate HD for a minimum of 12 weeks prior to Day 1. *CKD staging will be based on the five-stage system for classification of CKD based on KDIGO guidelines.
4. Hemodialysis patients with single-pool Kt/V ≥ 1.2 or urea reduction ratio ≥ 65%.

   *Single-pool Kt/V or urea reduction ratio will be based on results measured within 4 weeks prior to screening or during the screening period.
5. Patients must be on stable doses of IV injections of ESA (including biosimilars) for at least 6 weeks prior to Day 1.

   Minimum ESA dose;
   * Epoetin alfa, epoetin beta, and epoetin kappa: ≥1,500 U/week
   * Darbepoetin alfa: ≥20 µg/week
   * Mircera®: ≥30 µg/2 weeks
6. Mean of the 2 most recent local laboratory Hb screening values obtained at least 6 days apart, must be 9.0 g/dL to 12.0 g/dL, inclusive, with a difference of ≤1.5 g/dL between the highest and the lowest value.
7. Patients with serum ferritin ≥100 ng/mL at screening.
8. Patients with transferrin saturation (TSAT) ≥20% at screening.
9. Serum folate concentrations ≥lower limit of normal (LLN) at screening.
10. Serum total vitamin B12 concentrations ≥LLN at screening.

Exclusion Criteria:

1. Active acute or chronic infection, or uncontrolled or symptomatic inflammatory disease other than glomerulonephritis that could impact erythropoiesis (e.g., systemic lupus erythematosus, rheumatoid arthritis, celiac disease), or a C reactive protein level 40> mg/L (high sensitive C-reactive protein level > 10 mg/L).
2. By history or current clinical evidence, patients with active acute hepatitis B virus (HBV) or hepatitis C virus (HCV) infection should be excluded. Routine screening for HBV, HCV, and human immunodeficiency virus (HIV) infection is not required in this protocol. Chronic HBV/HCV infection with liver function tests (LFT) >3 times of normal are excluded. Known HIV positive patients are excluded.
3. History or clinical evidence of cardiovascular, hematologic, hepatic, or any physical conditions that, in the opinion of the Investigator, would compromise participation in the study.
4. Any of the following laboratory abnormalities at screening visit;

   * Alanine transaminase (ALT) >3 x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) >3 x ULN
   * Total bilirubin >1.5 x ULN
5. Chronic congestive heart failure (New York Heart Association class III or IV).
6. High risk for early withdrawal or interruption of the study (due to myocardial infarction, severe or unstable coronary artery disease, stroke, or severe liver disease) within the 12 weeks before Screening or during Screening.
7. Uncontrolled hypertension defined as a sitting systolic blood pressure ≥170 mmHg and/or diastolic blood pressure ≥100 mmHg.
8. History of active malignancy except for cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, or in situ cancer at any site.
9. Patients with a history of overt gastrointestinal bleeding or any other bleeding episode associated with a fall in Hb of ≥1 g/dL within the last 8 weeks prior to Screening.
10. Known history of myelodysplastic syndrome, multiple myeloma, hereditary hematologic disease such as thalassemia, sickle cell anemia, pure red cell aplasia, or other known causes for anemia other than CKD, hemosiderosis, hemochromatosis, known coagulation disorder, or hypercoagulable condition.
11. Any prior functioning organ transplant or a scheduled organ transplantation, or anephric state (one or both kidneys).
12. Planned elective surgery that could lead to significant blood loss during the study period.
13. Hypoalbuminemia (Serum albumin <2.5 g/dL) at Screening Visit.
14. Androgen, deferoxamine, deferiprone, or deferasirox therapy within 12 weeks prior to Day 1.
15. Life expectancy of <12 months.
16. Cognitive or psychiatric condition rendering the patient unable to be cooperative with and complete study requirements.
17. Hypersensitivity to any one of the investigational drugs or its excipients.
18. Received a blood transfusion (including RBC transfusion) within the 12 weeks prior to Screening, or blood transfusion is anticipated during the study period (excluding temporary blood transfusion given in case of blood loss due to accident or surgery).
19. Immunosuppressive therapy (tacrolimus/cyclosporine, and other than corticosteroids for a chronic condition) within 12 weeks prior to Day 1.
20. History of alcohol or drug abuse within the past 2 years and inability to avoid consumption of more than >3 alcoholic beverages per day.
21. Use of an investigational medication or treatment, participation in an investigational interventional study, or carryover effect of an investigational treatment expected during the study.
22. Females of childbearing potential or males who are unable/unwilling to take adequate contraceptive precautions defined by the protocol for the duration of the study and for at least 4 months for male subjects and 7 months for female patients after the end of the study. Females with a positive pregnancy test result within 24 hours prior to study entry, are otherwise known to be pregnant, plan to become pregnant in the next 12 months or are currently breastfeeding.
23. Patients who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or patients who are Sponsor or clinical research organization (CRO) employees directly involved in the conduct of the study.
24. Patients with very limited functional capacity for which a target Hb value of 12 g/dL may have a lower benefit/risk ratio.
25. Any medical condition (patients weighing over 150 kg) that, in the opinion of the Investigator, may pose a safety risk to a patient in this study, may confound efficacy or safety assessment, or may interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Mean change in hemoglobin (Hb) | Over Week 20 to Week 28
  Mean change from Baseline in Hb averaged over Week 20 to Week 28 without the use of rescue therapy (i.e., transfusion, or any approved ESA for all patients) within 6 weeks prior to and during the 8-week evaluation period.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Jeong Choi, Study Director — Genexine, Inc.
Locations (9):
- Georgia (4):
  - Batumi Dialysis and Nephrology Center, Batumi
  - Clinical Center for Nephrology Development, Tbilisi
  - L.Managadze National Center of Urology, Tbilisi
  - Tbilisi Heart And Vascular Clinic, Tbilisi
- South Korea (5):
  - Korea University Ansan Hospital, Ansan
  - St Mary's Incheon Hospital, Incheon
  - Kangdong KyungHee University Hospital, Seoul
  - St Mary's Seoul Hospital, Seoul
  - St Mary's Yeouido Hospital, Seoul